CLINICAL TRIAL: NCT06235801
Title: A Phase I/II Study of Gilteritinib and Momelotinib for Patients With Relapsed or Refractory FLT3-Mutated Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0438; NCI-2024-00669 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid | interventions — gilteritinib; N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Phase 1/Phase 2 (Experimental): Participants who are enrolled in Part 1, the dose of momelotinib you receive will depend on when you join this study. Participants you are enrolled in Part 2, you will receive momelotinib at the recommended dose that was found in Part 1. All participants will receive the same dose level of gilteritinib. Cycle 1 will be 35 days in length. Momelotinib will be administered once daily by mouth on days 1-35. Gilteritinib will be administered once daily by mouth on days 8-35. Cycles 2 and beyond will be 28 days in length. Momelotinib and gilteritinib will be administered once daily by mouth on days 1-28.
  Interventions: Drug: Gilteritinib; Drug: Momelotinib

INTERVENTIONS:
Drug: Gilteritinib — Given by PO
Drug: Momelotinib — Given by PO

SUMMARY:
To learn the recommended dose of momelotinib that can be given in combination with gilteritinib to participants with AML.

DETAILED DESCRIPTION:
Primary Objectives

* Phase I: To establish the minimum safe and biologically-effective dose of momelotinib in combination with gilteritinib in relapsed/refractory FLT3-mutated AML
* Phase II: To determine the modified CRc rate of the regimen, including complete remission (CR), CR with incomplete hematologic recovery (CRi) or morphologic leukemia free state (MLFS)

Secondary Objectives

* To assess other efficacy endpoints (CR rate, measurable residual disease negativity by flow cytometry and FLT3 PCR, relapse-free survival, overall survival)
* To assess proportion of participants proceeding to allogeneic hematopoietic stem cell transplantation
* To determine the safety of the combination regimen

Exploratory Objectives

* To evaluate the impact of baseline genomic alterations on response and survival of the combination regimen
* To determine the impact of baseline FLT3 allelic ratio on response and survival
* To evaluate the pharmacokinetics (e.g. AUC, Cmax, Tmax and half-life) of momelotinib in the combination regimen
* To evaluate changes in circulating cytokine levels in response to treatment
* To evaluate inhibition of FLT3 signaling and inhibition of JAK/STAT signaling pathways
* To evaluate other biomarkers associated with response and resistance to the combination regimen

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis:

   a) Adults ≥18 years with relapsed/refractory FLT3-mutated AML. Participants with either FLT3-ITD or FLT3 D835/D836 mutations will be eligible
2. Performance status ≤3 (ECOG Scale).
3. Adequate liver and renal function as defined by the following criteria:

   1. Total serum bilirubin ≤ 2 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the PI
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3 x ULN, unless due to the underlying leukemia approved by the PI

   d) Creatinine clearance ≥ 30 mL/min
4. Willingness to use adequate contraception prior to study entry, for the duration of study participation, and for 4 months after completion of study participation. For women of childbearing potential, adequate methods of contraception include: complete abstinence, hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal Ligation or hysterectomy, participants/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Congenital long QT syndrome or QTcF >450 msec. Repeat EKGs after correction of electrolytes or discontinuation of QT prolonging medications are allowed to meet entry criteria. In cases where QTcF >450 msec is considered to be falsely increased due to inaccurate automated reading and not clinically significant (e.g. due to bundle branch block), participants are still eligible if cardiologist reviews and documents that QTcF is ≤ 450 msec when manually measured.
2. Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment).
3. Active Class III-V cardiac failure as defined by the New York Heart Association Functional Classification.
4. Active central nervous system leukemia
5. Child-Turcotte-Pugh class C cirrhosis
6. Known human immunodeficiency virus (HIV) seropositive.
7. Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection Note: Participants who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Participants who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
8. Participants with a prior or concurrent malignancy whose natural history or treatment is not anticipated to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the PI
9. Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or participant has rapidly progressive disease judged to be life-threatening by the investigator.

   Prior recent treatment with corticosteroids, hydroxyurea and/or cytarabine (given for cytoreduction) permitted.
10. Inability to swallow
11. Unable or unwilling to sign informed consent
12. Pregnant women will not be eligible; A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: i. Is a woman of nonchildbearing potential (WONCBP), OR ii. Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, during the intervention period and for at least 4 month after the last dose of study drug.
13. Participants with psychiatric illness/social situations that would limit compliance with study requirements.
14. History of allergic reactions attributed to compounds of similar chemical or biologic composition to gilteritinib, momelotinib or other agents used in study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, MD, Principal Investigator — MD Anderson Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org